CLINICAL TRIAL: NCT01454141
Title: Cognitive Control Training for Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: BU-2182E
Record Dates: First submitted 2011-10-13; First posted 2011-10-18 (Estimated); Last update posted 2011-10-18 (Estimated); Status verified 2011-10

CONDITIONS: Depression
Keywords: Depressed mood
MeSH Terms: conditions — Depression; Consciousness Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Peripheral Vision Task (Experimental): During this task participants viewed a circular array of 15 discs and were asked to move their attention, but not their eyes, clockwise around the array while auditory tones were presented. Following the presentation of a distinct target tone, the discs changed color and participants reported the color of the disc by pressing a designated button on the keyboard. This task was developed to be a non-active control condition, targeting visual and occipital areas of the brain, and therefore allows us to discriminate between the effects of completing a computer-based task from interventions that specifically target the PFC.
  Interventions: Other: Peripheral Vision Task
- Cognitive Control Training (Experimental): Cognitive Control Training (CCT) A modified version of the Paced Auditory Serial Addition Task (PASAT) and the Attention Control Intervention were used to train participants' attentional control in accordance with procedures used by Siegle and colleagues.
  Interventions: Other: Cognitive Control Training

INTERVENTIONS:
Other: Cognitive Control Training — Three sessions of CCT.
  Arms: Cognitive Control Training
Other: Peripheral Vision Task — Three sessions of PVT.
  Arms: Peripheral Vision Task

SUMMARY:
Depression is frequently characterized by patterns of inflexible, maladaptive, and ruminative thinking styles; these patterns themselves are thought to result from a combination of decreased attentional control, decreased executive functioning, and increased negative affect. Specifically, the dorsolateral prefrontal cortex has been hypothesized to play a central role in emotion regulation by recruiting resources necessary for executive control. Recent advances have been made in neurobehavioral training strategies as interventions for emotional disorders such as depression. Cognitive control training (CCT) uses computer-based exercises to recruit and activate prefrontal neural networks via repeated behavioral exercises, with the aim of strengthening cognitive and emotional functions. A previous study found that severely depressed participants who received CCT exhibited reduced negative affect and rumination as well as improved focus and concentration. The present study aimed to extend this line of research by employing a more stringent control group and testing the efficacy of three sessions of CCT over a two-week period in a community population with depressed mood. Forty-eight participants with high BDI-II scores were randomized to CCT or a comparison condition (Peripheral Vision Training; PVT). The investigators hypothesized that relative to a control condition (PVT), CCT would be associated with less self-reported negative mood and emotional reactivity.

ELIGIBILITY:
Inclusion Criteria:

* BU students and local community members.
* At least 18 years of age.
* Familiarity with a computer keyboard.
* BDI-II score ≥ 17

Exclusion Criteria:

* BDI-II score < 17, or > 35

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2010-07; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Change in Beck Depression Inventory | two weeks
  Change score in BDI was assessed between CCT and PVT groups.

SECONDARY OUTCOMES:
Change in Positive and Negative Affective Scale (PANAS) | two weeks
  We looked at the change scores in positive and negative affectivity between CCT and PVT groups.
Emotional Response and Recovery Task | two weeks
  We looked at the emotional responses to IAPS images between CCT and PVT groups.
Changes in Visual Analog Scales | two weeks
  We looked at the change scores in visual analog scales (happy/sad) between CCT and PVT groups.

CONTACTS AND LOCATIONS:
Locations (1):
- Boston University, Boston, Massachusetts, United States